CLINICAL TRIAL: NCT00990522
Title: A Prospective, Randomized, Controlled Study of the Efficacy of Sharp Debridement for the Management of Chronic Wounds
Brief Title: Study of the Efficacy of Sharp Debridement for the Management of Chronic Wounds
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled, per PI discretion
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Prinicipal Investigator, Southwest Regional Wound Care Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 56-RW-014
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Wounds
Keywords: sharp debridment; patients with full thickness wounds of greater than 30 days duration
MeSH Terms: conditions — Wounds and Injuries | interventions — Debridement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- debridement (Experimental): monthly vs weekly debridement
  Interventions: Procedure: debridement

INTERVENTIONS:
Procedure: debridement — There will be two (2) subject groups in the study. Subjects will be randomized into either the monthly debridement group or the weekly debridement group.

SUMMARY:
Standard care of care and up to twelve (12) weekly debridements. Subjects randomized into the weekly debridement group will receive up to twelve (12) debridement during the twelve (12) weeks of the study. There will be two (2) subject groups in the study. Subjects will be randomized into either the monthly debridement group or the weekly debridement group.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate subjects enrolled and randomized to the weekly sharp debridement group.

The major secondary objectives are incidence of complete wound closure at Week 12, rate of healing, ulcer recurrence, wound characteristics, and microbiologic information.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have evidence of a full-thickness cutaneous wound of at least 30 days duration.
2. Subject must be at least 18 years of age.
3. Subject must have a minimum life expectancy of at least 1 year to be determined by the Investigator.
4. The study ulcer must be from 1 cm2 to 20 cm2 in size.
5. The study ulcer must have been present for at least 30 days at study Day -7.
6. The subject's Glycosylated hemoglobin (HbA1C) must be equal to or less than 10.0% for subjects with diagnosed diabetes at study Day 0.
7. The subject, legal guardian or authorized representative must have understood, signed and dated the IRB approved informed consent form.
8. The subject must be available for evaluation on a weekly basis for the twelve (12) weeks of the study. Visits at Week 13 and Week 14 are required for initial wound healing, which is achieved in study Week 11 or 12. The Investigator will evaluate both groups at Week 16. Subjects must be available for evaluation at Week 16.
9. The subject's TCpO2 must be equal to or greater than 25 mm of mercury in the periwound area and ABI greater than 0.7.

Exclusion Criteria:

1. Subject whose ulcer has healed 30% or greater from the evaluation Study day -7 to the post-debridement Study Day 0 as determined by wound measurements using ARANZ Silhouette
2. A history of alcohol or substance abuse, within the previous year, which could, or in the judgment of the Investigator, would interfere with study compliance or protocol requirements.
3. Participation in clinical trials evaluating investigational pharmaceuticals, biologics or devices within 30 days of admission to the study.
4. Subject with a history of receiving any of the following within the last 30 days: systemic corticosteroids exceeding a total daily dose of 20mg, immunosuppressive agents, radiation therapy or chemotherapy. Anticipated use of the above during the study period will also exclude a subject from entry into the study. Topical and inhaled corticosteroids are not prohibited.
5. Subjects with medical comorbidities known to affect wound healing such as end stage renal disease, severe hepatic insufficiency, vasculitis, and HIV will be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate subjects enrolled and randomized to the weekly sharp debridement group. | 12 weeks

SECONDARY OUTCOMES:
The major secondary objectives are incidence of complete wound closure at Week 12, rate of healing, ulcer recurrence, wound characteristics, and microbiologic information. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Randall Wolcott, M.D., Principal Investigator — Southwest Regional Wound Care Center